CLINICAL TRIAL: NCT05330403
Title: The Moxibustion-Induced Thermal Transport Effect Between The Heart And Lung Meridians With Infrared Thermography
Brief Title: The Moxibustion-Induced Thermal Transport Effect Between The Heart And Lung Meridians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019ZY010-MERIDIAN
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Meridians
Keywords: heart and lung meridians; site specificity; infrared thermography; moxibustion; thermal transport
MeSH Terms: interventions — Moxibustion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the lung meridian intervention group (Experimental): moxibustion intervention was performed over Site 1 (LU5) of the lung meridian
  Interventions: Procedure: Moxibustion
- the heart meridian intervention group (Experimental): moxibustion intervention was applied over Site 4 (HT3) of the heart meridian
  Interventions: Procedure: Moxibustion

INTERVENTIONS:
Procedure: Moxibustion — In this study, suspended moxibustion was performed by holding an ignited moxa stick at a certain distance (about 3-4 cm) over the skin surface, keeping the moxibustion Site warm without burning the skin.
  In the heart meridian intervention group, moxibustion was applied over Site 4 (HT3) of the heart meridian.
  In the lung meridian intervention group, moxibustion was performed over Site 1 (LU5) of the lung meridian.

SUMMARY:
Although some important progresses were made in the field of the meridian research, no breakthroughs have been achieved. Besides,there are some problems in meridian researches. Particularly, previous research of meridian phenomenon involved lots of subjective elements and outcomes. Researches that use modern scientific techniques to investigate the biological characteristics of meridian phenomenon are urgently needed. Therefore, this study was designed to assess the heat transport characteristics of meridian phenomenon for the Heart and Lung meridians by using infrared thermography. Thus, the biological characteristics of meridian phenomenon could be presented objectively in a scientific methodology.

DETAILED DESCRIPTION:
80 eligible subjects were finally included. Among them, 40 participants were assigned to the lung meridian intervention group, and 40 participants were assigned to the heart meridian intervention group. All 80 participants completed the trial.

ELIGIBILITY:
Inclusion Criteria:

* Had recent medical examination records confirming the absence of cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological diseases
* 20 ≤ age ≤ 40 years, male or female
* Had the ability to communicate with others normally
* An understanding of the entire study protocol
* Signed written informed consent

Exclusion Criteria:

* Had mental illnesses, severe depression, alcohol dependence or a history of drug abuse
* Pregnant or lactating
* Were participating in other trials

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Temperature change of relevant sites | Baseline, Moxibustion 5 min, Moxibustion 10 min, Moxibustion 15 min, 5 minutes after stopping moxibustion
  Infrared thermal imaging was used to record baseline temperature and the temperature change of corresponding sites along the Heart and Lung meridians.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Jiang Y, Hu H, Lou J, Zhang Y, He X, Wu Y, Fang J, Shao X, Fang J. The Moxibustion-Induced Thermal Transport Effect Between the Heart and Lung Meridians With Infrared Thermography. Front Cardiovasc Med. 2022 May 13;9:817901. doi: 10.3389/fcvm.2022.817901. eCollection 2022. PMID 35647050